CLINICAL TRIAL: NCT01809873
Title: Sustainable Financial Incentives To Improve Prescription Practices For Malaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Moi University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Health Services Research
Other Study IDs: Pro00035154
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Malaria
Keywords: Malaria; Diagnostics; Health Services
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Performance based incentives (Experimental): Performance based incentives: The Incentive arm will receive monthly visits and external quality assurance of malaria diagnostic accuracy, identical to the comparison. Incentive arm will also receive quarterly incentives linked to performance of the facility around six indicators of appropriate malaria case management
  Interventions: Behavioral: Performance based incentives
- Comparison (No Intervention): The comparison arm will receive monthly visits and monthly external quality assurance of malaria diagnostic accuracy.

INTERVENTIONS:
Behavioral: Performance based incentives — Facilities enrolled in the intervention arm will receive a financial incentive that is based on their diagnosis and prescription practices for malaria over that quarter. The intervention will last 12 months.
  Arms: Performance based incentives

SUMMARY:
This project aims to test an innovative, sustainable financial incentive designed to reduce the number of non-malarial fevers that are treated inappropriately with antimalarial drugs.

DETAILED DESCRIPTION:
Global investments in controlling malaria have led to some exciting reductions in the burden of malaria. In some areas, malaria-related deaths have dropped by more than 90%. As malaria transmission declines, a greater fraction of pediatric fevers are from other causes. However, these fevers continue to be treated as malaria, often despite the availability of diagnostic testing. In a typical rural health facility in Kenya, more than 90% of febrile patients are prescribed an antimalarial when no diagnostic tests are available. Even when microscopy or rapid diagnostic tests (RDTs) are available, between 50-80% of patients with a negative test are nonetheless prescribed antimalarials. Inappropriately treated fevers in children can lead to serious consequences for the patient and can accelerate the spread of drug resistance. In addition to the risk to patients, overuse of antimalarials also puts a financial strain on the government health system. Although there is considerable incentive for governments to reduce drug costs and wastage, the financial pressure is not experienced at the appropriate levels of decision-making.

This project aims to test an innovative, sustainable financial incentive designed to reduce the number of non-malarial fevers that are treated inappropriately with antimalarial drugs. The study team will test a financial incentive targeted at the health facility to determine if it improves adherence to diagnostic results and clinical protocols. Eighteen rural health facilities in Western Kenya will be enrolled and randomly allocated to one of two arms. The study team will compare the effectiveness of clinical and technical training in diagnosis of malaria alone (Arm 1) to training plus financial incentives linked to prescription practices (Arm 2) in improving diagnosis and treatment of malaria and non-malaria fevers. The practice of prescribing antimalarials to patients with a negative diagnostic will be compared between facilities with and without the incentive structure. Secondary outcomes will include sensitivity and specificity of routine microscopy at health centers, use of alternative treatments for slide negative fevers, and frequency of stock-outs of antimalarial drugs.

This project will tackle an important implementation research problem. It seeks to test solutions to the problem of poor adherence to evidence-based clinical guidelines for malaria treatment, and thereby reduce inappropriate antimalarial drug use and drug wastage. This project will be conducted in collaboration with Kenya's Division of Malaria Control and avenues to roll-out the intervention, if successful, will be actively explored.

ELIGIBILITY:
Inclusion Criteria:

* Health facility (level 3) in Western or Rift valley province, within the Academic Model Providing Access to Healthcare (AMPATH) catchment area
* Consent from Provincial Medical Officer of Health, District Medical Officer of Health and Health facility in-charge
* Functioning laboratory including microscopic diagnosis of malaria and at least one laboratory technician.

Exclusion Criteria:

* Lack of consent from any level
* Lack of adequate laboratory infrastructure or personnel

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14862 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Proportion of children under 5 years of age who are treated with antimalarials following a negative malaria test | At one year post-intervention
  The study is designed to detect a reduction in the proportion of children under 5 years of age who are prescribed antimalarials following a negative malaria diagnostic test between the intervention and comparison arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Moi University, Eldoret, Rift Valley Province, Kenya

REFERENCES:
- [Derived] Menya D, Platt A, Manji I, Sang E, Wafula R, Ren J, Cheruiyot O, Armstrong J, Neelon B, O'Meara WP. Using pay for performance incentives (P4P) to improve management of suspected malaria fevers in rural Kenya: a cluster randomized controlled trial. BMC Med. 2015 Oct 16;13:268. doi: 10.1186/s12916-015-0497-y. PMID 26472130
- [Derived] Menya D, Logedi J, Manji I, Armstrong J, Neelon B, O'Meara WP. An innovative pay-for-performance (P4P) strategy for improving malaria management in rural Kenya: protocol for a cluster randomized controlled trial. Implement Sci. 2013 May 8;8:48. doi: 10.1186/1748-5908-8-48. PMID 23656836